CLINICAL TRIAL: NCT02593981
Title: To Sleep, Perchance to Dream: A Randomized, Placebo-Controlled Study to Test a Fruit/Honey-Based Foodstuff for Sleep Problems in Older Adults
Brief Title: Addressing Sleep Problems in Older Adults
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to obtain study agent
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Brent A. Bauer, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-006031
Record Dates: First submitted 2015-10-29; First posted 2015-11-02 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Sleep
Keywords: sleep; fruit; honey; geriatric
MeSH Terms: interventions — Fruit

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fruit/Honey Drink (Active Comparator): Fruit/Honey Drink (2 canisters) will be taken orally twice a day. Subjects will consume the drink on days 1 through 28.
  Interventions: Dietary Supplement: Fruit/Honey drink
- Placebo (Placebo Comparator): Placebo (2 canisters) will be taken orally twice a day. Subjects will consume the placebo drink on days 1 through 28.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Fruit/Honey drink — 2 canisters of powder containing fruit/honey mix to be mixed with water and ingested twice a day for 28 days
  Arms: Fruit/Honey Drink
Dietary Supplement: Placebo — 2 canisters of Placebo powder containing non-active ingredient to be mixed with water and ingested twice a day for 28 days
  Arms: Placebo

SUMMARY:
As many as 57% of older adults complain of major disruption of sleep, 29% struggle to fall asleep and 19% complain of early-morning awakening. The implications of this sleep deprivation are sobering, particularly among older individuals.

The primary goal of this study is to determine whether a palatable foodstuff which contains a fruit/honey drink and which is taken every evening before bedtime leads to improved sleep in community-living individuals with sleep problems.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled double-blinded pilot study to explore the use of a fruit/honey drink product for improving sleep in older adults. The purpose of this study is to estimate the effects of a fruit/honey drink using various assessment tools when used as short-term intervention.

This trial proposes to enroll a total of 60 community based older adults. All study patients will be instructed to take the study product every day for 28 days. During which time, study subjects will return weekly to complete study visits for a total of 4 visits.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 60 years old at the time of study registration.
2. Individual describes trouble either falling asleep or staying asleep at study entry.
3. Willing to participate in all aspects of the study.
4. Willing to avoid kiwifruit, cherry, and honey for 4 weeks while on this study.
5. Willing to avoid changes to current sleep medications (may use a stable dose of a currently prescribe sleep medication during the first 4 weeks after stating the intervention).

Exclusion Criteria:

1. Allergic to kiwifruit, cherries, honey, apples, or bananas.
2. Hospitalized or living in a care facility at the time of enrollment.
3. Clinical evidence of active malignant disease (cancer), as per healthcare provider's clinical judgment.
4. Any cancer therapy (for example, chemotherapy, hormonal therapy, radiation, surgery, immunotherapy) in the preceding 3 months.
5. Healthcare provider does not think that study candidate has a specific health problem that precludes participation.
6. Allergy or intolerance of milk products.
7. Women of child bearing potential.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03 (Estimated); Primary Completion 2019-02 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
PSQI score | 28 days
  Pittsburgh Sleep Quality Index (PSQI):

CONTACTS AND LOCATIONS:
Overall Officials: Brent Bauer, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No